CLINICAL TRIAL: NCT04231643
Title: A Randomized, Controlled Trial of Cannabis in Bipolar Disorder Patients and Healthy Volunteers Evaluating Cognition and Endocannabinoid Levels
Brief Title: Effects of Cannabis on Cognition and Endocannabinoid Levels in Bipolar Disorder Patients and Healthy Volunteers
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Budgetary limitations prevented us from completing our planned sample size.
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, William Perry, Professor in Residence of Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 180356; R01DA043535 (NIH)
Record Dates: First submitted 2020-01-08; First posted 2020-01-18 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Bipolar Disorder
Keywords: cannabidiol; THC
MeSH Terms: conditions — Bipolar Disorder | interventions — Dronabinol; Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bipolar Disorder (Experimental): adults with bipolar disorder
  Interventions: Drug: Dronabinol; Drug: Epidiolex; Drug: Placebos
- Healthy Volunteers (Active Comparator): adults with no psychiatric disease
  Interventions: Drug: Dronabinol; Drug: Epidiolex; Drug: Placebos

INTERVENTIONS:
Drug: Dronabinol — one-time oral administration of 5 mg dronabinol
Drug: Epidiolex — one-time oral administration of 600 mg Epidiolex
Drug: Placebos — one-time oral administration of placebo

SUMMARY:
Cannabis use is associated with younger age at onset of bipolar disorder, poor outcome, and more frequent manic episodes, but the effects of cannabis on cognition are less clear. Contrary to reports among non-psychiatric patients, cannabis may improve cognition among people with bipolar disorder. Nevertheless, no study to date has systematically tested the acute effects of cannabis on cognition in bipolar disorder. Therefore, the investigators propose to determine the effects of oral cannabinoid administration on cognitive domains relevant to bipolar disorder, e.g., arousal, decision making, cognitive control, inhibition, and temporal perception (sense of timing). In addition, the investigators will evaluate different doses of the two major components of cannabis, cannabidiol and ∆9-tetrahydrocannabinol, and compare them to placebo on these neurocognitive measures. The investigators will also test the effects of acute exposure to cannabinoids on cerebrospinal levels of anandamide and homovanillic acid - markers of endocannabinoid and dopamine activity in the brain, respectively. These studies will provide information that effectively bridges the fields of addiction and general psychiatry, informing treatment development for co-morbid substance abuse and psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

1. For subjects in BD group, DSM-5 criteria for Bipolar Disorder as determined by the Structured Clinical Interview for DSM-5 (SCID).
2. Young Mania Rating Scale (YMRS) < 12.
3. Infrequent cannabis use as defined by a history of cannabis use and current use no more than 4 times per month.
4. Willing to abstain from cannabis use for at least two days prior to the experimental visit.

Exclusion Criteria:

1. Hamilton Depression Rating Scale (HDRS) score > 10.
2. Suicidality. Exposure to cannabis does not lead to depression but it may be associated with suicidal thoughts and attempts. Therefore, the Center for Epidemiological Studies-Depression Scale (CES-D) subscale measuring suicidal ideation ("I wished I were dead". "I wanted to hurt myself") will be completed. Should any of these items be answered affirmatively, e.g., the subject has endorsed these items for at least 1-2 days in the last week, the subject will not be enrolled in the study.
3. The Substance Abuse Module of the Diagnostic Interview Schedule for DSM-5 will be administered to exclude individuals with current substance use disorders.
4. Clinically significant or unstable medical condition. Subjects will undergo a medical evaluation (H&P, toxicology screening, and for females of childbearing potential, pregnancy testing (utilizing a human chorionic gonadotropin (hCG) urine test). Individuals with significant cardiovascular disease (e.g., angina, myocardial infarction or stroke), hepatic or renal disease, uncontrolled hypertension, and chronic pulmonary disease (e.g., asthma, COPD), will be excluded. With respect to cardiovascular and pulmonary status, a clinician will screen participants with a tool developed for this purpose (Appendix 3 Cardiopulmonary Screen). Hepatic and renal disease will be evaluated with liver and renal function laboratory tests. Females who are pregnant or lactating will be excluded.
5. Infections - evidence of skin infection at lumbar puncture site.
6. To avoid confounding of cognitive testing, a neurological disorder such as seizures, stroke, Parkinson's disease, dementia, or a history of head injury with loss of consciousness for at least 15 minutes will be excluded.
7. Unwilling to refrain from driving or operate heavy machinery for four hours after consuming study medication. This criterion is consistent with current expert recommendations on driving following the use of cannabis.
8. Additionally, because the hBPM paradigm requires participants to be ambulatory, those who cannot ambulate independently (e.g., require a wheelchair) or those who have a motor disease (e.g., multiple sclerosis, cerebral palsy) will be excluded.
9. A previous adverse reaction to cannabinoids will be cause for exclusion as will a historical diagnosis of cannabis use disorder.
10. Positive result on Draeger 5000 test indicating recent cannabis use.
11. Unwillingness to prevent pregnancy during the cannabinoid administration portion of the study (using birth control in female participants of child-bearing age) Acceptable methods of birth control are: oral contraceptive pills, diaphragm, condom, progestin implant, intrauterine contraceptive device, sterilization, etc.
12. Any active opportunistic infection or malignant condition requiring acute treatment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants will be asked about which gender they identify with
Enrollment: 19 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Score on Iowa Gambling Task | one day
  This is an experimental measure and not a scale with specific anchor points. Lower scores reflect increased risk-taking
Score on Progressive Ratio Test | one day
  This is an experimental measure and not a scale with specific anchor points. Higher scores indicate increased willingness to work for a reward
Scores on Probabilistic Learning Task | one day
  This is an experimental measure and not a scale with specific anchor points. Measures decision-making strategies such as win-stay, lose-shift.
Scores on Continuous Performance Task | one day
  This is an experimental measure and not a scale with specific anchor points. Higher scores reflect better attention and ability to discriminate important information from unimportant information
Percent Prepulse Inhibition (PPI) | one day
  This is a physiological measure and not a scale with specific anchor points. Higher percent PPI reflects better sensorimotor gating
motor activity in the human Behavioral Pattern Monitor | one day
  This is an experimental measure and not a scale with specific anchor points. Subjects' behavior in an open field (a room filled with novel objects) is quantified over a 15-minute period via amount of motor activity as measured by a wearable accelerometer. Increased motor activity reflects increased tendency to engage in exploratory behavior.
object interactions in the human Behavioral Pattern Monitor | one day
  This is an experimental measure and not a scale with specific anchor points. Subjects' behavior in an open field (a room filled with novel objects) is quantified over a 15-minute period via video ratings that quantify number of interactions with novel objects. Increased object interactions reflects increased novelty-seeking behavior.
cerebrospinal fluid levels of anandamide | one day
  Reflects increased availability of the endogenous cannabinoid anandamide in the brain

CONTACTS AND LOCATIONS:
Overall Officials: William Perry, PhD, Principal Investigator — UCSD
Locations (1):
- UC San Diego Medical Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT04231643/ICF_000.pdf